CLINICAL TRIAL: NCT04954703
Title: Effects of Myofascial Release of IT Band With or Without Muscle Energy Technique of Gluteus Maximus and Tensor Fascia Lata With Iliotibial Band Syndrome.
Brief Title: Myofascial Release With and Without METS of Gluteus Maximus and Tensor Fascia Lata in ITB Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0104/Aqsa
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Iliotibial Band Syndrome
Keywords: ITB syndrome; Muscle energy technique (METS); Myofascial release
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle energy technique of gluteus maximus and tensor fascia lata (Experimental): INTERVENTIONAL GROUP (muscle energy technique of gluteus maximus and tensor fascia lata)
  Interventions: Other: Muscle energy technique of gluteus maximus and tensor fascia lata
- Myofascial release of iliotibial band (Active Comparator): CONTROL GROUP(Myofascial release of iliotibial band)
  Interventions: Other: Myofascial release of iliotibial band syndrome

INTERVENTIONS:
Other: Muscle energy technique of gluteus maximus and tensor fascia lata — it is used for lengthening of hypertonic muscles for relief of pain and range of motion.Position of patient is supine lying and therapist is at side of table .The patient leg is fully adducted to stretch IT band and then patient attempts to abduct the leg against resistance contracting the muscles being stretched at approximately 25% of maximum effort for 10 seconds. They then relax and the therapist lengthen it.
  Arms: Muscle energy technique of gluteus maximus and tensor fascia lata
Other: Myofascial release of iliotibial band syndrome — Myofascial release of IT band Syndrome. Therapist fingers track up and down your ITB with fingertips to find the most tender spots and use a tennis ball to apply small, circular, light release in those places.
  Arms: Myofascial release of iliotibial band

SUMMARY:
This Study Will Be Conducted to Evaluate the Effects Of myofascial release of IT band with or without muscle energy technique of gluteus maximus and tensor fascia Lata with iliotibial band syndrome. Data Will Be Collected from Haider memorial hospital in Vehari. Study will include 24 patients of both genders with pain on lateral side of pain confirmed by positive ober test. Treatment group patient will receive myofascial release and muscle energy technique of gluteus maximus & tensor fascia Lata muscle to relieve pain of IT band syndrome while control group will only receive myofascial release treatment. All 24 patients will be stable during the study period. Study will be conducted based on 06 month time period after approval of synopsis. Patients will be studied and fill out questionnaire. All possible patients with iliotibial tract syndrome will be taken using consecutive sampling. Informed consent will be taken from all recruited patients. The results of this study will help to manage the pain of iliotibial tract & will be a randomized controlled trial

DETAILED DESCRIPTION:
The iliotibial tract is a dense fibrous connective tissue thickening of the fascia Lata on lateral side of the thigh. The ITB is attached proximally at the greater trochanter of femur with fascial involvement of the tensor fascia Lata and the gluteus maximus and gluteus Medius muscles to lateral condyle of tibia. The most common injury of lateral knee is iliotibial band syndrome(ITBS). ITBS is an overuse injury results from repetitive friction of the iliotibial band (ITB) over the lateral femoral epicondyle, biomechanical studies explained that a maximal zone of impingement is at approximately 30° of knee flexion. Prevalence of ITBS accounts for 15% to 24% in all overuse injuries in non-experimental investigations. Epidemiologic studies demonstrates ITBS as the most common cause of lateral knee symptoms with a reported incidence ranging from 1.6% to 12%.

ITBS is an overuse injury from repetitive movements cause friction, irritation, and pain when moving the knee joint. Prospective research demonstrate that the greater internal rotation at the knee joint and increased adduction angles of the hip joint play important role in the etiology of ITBS and that the strain rate in the iliotibial bands is greater in persons with repetitive movements of knee joints compared to other persons.

Presentation of Iliotibial band syndrome is increased knee internal rotation, decreased rear foot eversion, tibial internal rotation and hip adduction angles at heel strike with maximum internal rotation at the knee and decreased total abduction and adduction range of motion at the hip during stance phase during stance. It also exhibits greater invertor moments at their feet, decreased abduction and flexion at their hip joint and to reach maximum hip flexion angles earlier than healthy individuals. female gender may be a predisposing factor of iliotibial band syndrome. Iliotibial band friction syndrome is an overuse injury mostly seen in long distance runners, cyclists, and military personnel with estimated incidence of 1.6%-52% .ITB length is measured by Ober's test and modified Ober's test, with hip adduction angle that is monitored by using a fluid goniometer.

Manual therapy is first choice in treatment of ITBS consists of soft tissue release and medial patella mobilizations for relieve of pain and lengthening the ITB. Myofascial release with use of foam roller as a myofascial release tool is used to break up soft-tissue adhesions in the ITB . Studies also showed that myofascial release is beneficial for relieving lateral knee pain. With progression of patient performing the stretching regimen without pain, strengthening is also added to the rehabilitation program. Physical Interventions such static stretching, strengthening, manual therapy and neuromuscular re-education and muscle energy techniques are performed for treatment of ITBS. Active Release Technique and Myofascial Release Technique are also effective in patients with musculoskeletal pain but researches revealed that Myofascial Release Technique demonstrated has better outcomes than Active Release Technique in the management of Chronic pain.

The increased tone of gluteus maximus can be corrected with active pump techniques, combining of soft tissue mobilization with muscle energy techniques. Isometric of hip abduction and adduction strengthening also performed for relieve and gain range of motion in ITBS. MET is a treatment technique includes a willful constriction of a subject's muscle in a controlled bearing, against a counterforce that is given by the specialist. MET is utilized to diminish the pain, extend the tight muscles and belts, decrease muscle tone, enhances nearby flow, strengthen the feeble musculature, and mobilizes the joint restrictions. MET increase the extensibility of muscles and spinal range of motion, treating patients with reduced mobility. Muscle energy techniques involve post isometric relaxation and post facilitation stretching techniques. METS of specific muscles are used for improvement the efficacy of neurodynamic and lymphatic system

ELIGIBILITY:
Inclusion Criteria:

* patient having pain on lateral side of knee with positive ober's test

Exclusion Criteria:

* medically unstable patients
* others causes of lateral knee pain like meniscus and ligaments tear
* trauma causes
* other pathological condition of knee

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale | 3 weeks
  It is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
lower extremity functional scale | 3 weeks
  lower extremity functional scale score = sum (points for all 20 activities) Interpretation: Minimum score: 0 Maximum score: 80 The lower the score the greater the disability. The Minimal Detectable Change (MDC) is 9 scale points. The Minimal clinically Important Difference (MCID) is 9 scale points

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sana ullah, Principal Investigator — Riphah International University
Locations (1):
- Haider memorial hospital, Burewala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khaund R, Flynn SH. Iliotibial band syndrome: a common source of knee pain. Am Fam Physician. 2005 Apr 15;71(8):1545-50. PMID 15864895
- [Background] Holzer M, Padberg F. Intermittent theta burst stimulation (iTBS) ameliorates therapy-resistant depression: a case series. Brain Stimul. 2010 Jul;3(3):181-3. doi: 10.1016/j.brs.2009.10.004. Epub 2009 Nov 1. No abstract available. PMID 20633448
- [Background] De Maeseneer M, Boulet C, Willekens I, Lenchik L, De Mey J, Cattrysse E, Shahabpour M. Segond fracture: involvement of the iliotibial band, anterolateral ligament, and anterior arm of the biceps femoris in knee trauma. Skeletal Radiol. 2015 Mar;44(3):413-21. doi: 10.1007/s00256-014-2044-x. Epub 2014 Dec 4. PMID 25468067
- [Background] Subotnick SI. Limb length discrepancies of the lower extremity (the short leg syndrome). J Orthop Sports Phys Ther. 1981;3(1):11-6. doi: 10.2519/jospt.1981.3.1.11. PMID 18810144
- [Background] Fredericson M, Wolf C. Iliotibial band syndrome in runners: innovations in treatment. Sports Med. 2005;35(5):451-9. doi: 10.2165/00007256-200535050-00006. PMID 15896092